CLINICAL TRIAL: NCT02014285
Title: Muscle Ultrasound Signifies Condition Upgrade Leading Approach to Recovery
Acronym: MUSCULAR
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 00022113
Record Dates: First submitted 2013-11-27; First posted 2013-12-18 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-08

CONDITIONS: Acute Respiratory Failure; Critical Illness
Keywords: Acute Respiratory Failure; Critical Illness; Mechanical Ventilation; Muscle Architecture; Muscle Ultrasound
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Muscle tissue and serum/plasm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Muscle Ultrasound/Sample: 30 subjects enrolled from Wake Forest Baptist Health Intensive Care Units. Each study subject will undergo an ultrasound to examine the size and echogenicity of their muscles and a muscle biopsy from the rectus femoris. The muscles studied will include the biceps brachii, wrist extensors, quadriceps, and tibialis anterior.
  Interventions: Procedure: Muscle Ultrasound and Muscle Sample

INTERVENTIONS:
Procedure: Muscle Ultrasound and Muscle Sample — The muscles to undergo ultrasound will include the biceps brachii, wrist extensors, quadriceps, and tibialis anterior. A muscle sample will be taken from the rectus femoris.

SUMMARY:
Examination of serial muscle ultrasounds and muscle sampling within the population of ICU patients who require mechanical ventilation for acute respiratory failure, will lead to the ability of investigators to link specific baseline comorbidities, drugs, or fluid administrations, to the onset and duration of architectural changes within muscle and correlate ultimately with muscle function. With this study, we will be better able to understand the relationships between the pattern of resolution of the muscle architectural abnormalities within the context of multiple other clinical abnormalities and therapies present and rendered to ICU patients.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) is an extremely variable and heterogeneous syndrome that can be defined as an acute cardiopulmonary dysfunction requiring emergent artificial ventilation support. For patients with ARF, the mortality rate is higher than the general ICU mortality, with estimates ranging from 15-40% depending on the subgroups evaluated. In the largest, most recent report on ARF, the in-ICU mortality was 31% and the overall in-hospital mortality rate was 37%. Muscle weakness is an independent risk factor for mortality from ARF and contributes to long-term reductions in physical function in survivors. Muscle ultrasounds are non-invasive, quick and reproducible. They provide the opportunity of ICU staff to create a patient-specific exercise prescription based on both functional assessments and importantly the degree of muscle architecture abnormality detected by ultrasound. Serial examination of muscle ultrasound images obtained in mechanically ventilated acute respiratory failure patients will allow for better understanding of the time course of specific muscles' architectural abnormalities and the resolution of such abnormalities within hospital survivors. With this study, we will be better able to understand the relationships between the pattern of resolution of the muscle architectural abnormalities within the context of multiple other clinical abnormalities and therapies present and rendered to ICU patients. Muscle sampling used in conjunction with ultrasound in patients with ARF will allow for further characterization of the extent of and mechanisms underlying ARF induced muscle dysfunction in these patients. Furthermore, ultrasound guided muscle sampling allows this procedure to be done in a more efficient and effective manner. Study participants will consist of 30 patients with ARF admitted to the Intensive Care Units of Wake Forest University Baptist Medical Center. Muscle ultrasounds will occur at study enrollment and weekly thereafter, and will also include one imaging session as close to hospital discharge as possible. Muscle sampling will occur within 5 days of consent and approximately 2 months later. Handgrip strength, dynamometer, and physical performance tests will also be administered at ICU & hospital discharge and at 2 months post enrollment. The primary outcome will be to investigate the possibility of a relationship between the ultrasound data, muscle sample data, and functional measurements (length of stay, grip strength, SPPB, dynamometer, MRC, simultaneously accounting for severity of illness [APACHE III]).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mechanically ventilated via an endotracheal tube or mask
* New diagnosis of Acute Lung Injury or Sepsis

Exclusion Criteria:

* Upon Principle Investigator discretion, patient not suitable for study
* Moribund
* Other Research Study without co-enrollment permissions
* Pregnancy
* Primary neuropathies
* Amputees
* Inability to walk without assistance prior to diagnosis (use of cane or walker not exclusion)
* Preadmission immunocompromised state (HIV, >20mg prednisone/day, other immunosuppressive therapy)
* BMI >45 (difficulty obtaining biopsy)
* Underlying neuromuscular disease
* Acute stroke
* Hip fracture, unstable C spine, or pathological fracture
* Current hospitalization or transferring hospital stay >80 hours
* CPR previous to consent without signs of full neurologic recovery
* Previous hospitalization within past 30 days
* Cognitive impairment prior to ICU illness
* Re-admission to ICU within current admission
* Cancer therapy within the last 12 months
* Full dose anticoagulation therapy
* Known platelet count <100,000
* Known INR >1.5
* Known aPTT >1.5 upper limit of normal
* Patient on antiplatelet therapy (daily aspirin therapy is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will consist of 30 patients with Acute Respiratory Failure admitted to the Intensive Care Units of Wake Forest Baptist Health.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-11; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Days of Hospitalization | 2 months
  The ultrasound data analysis may allow for a correlation to be drawn between a pattern of ultrasound changes and length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Clark Files, MD, Principal Investigator — Wake Forest University Health Sciences; Peter E Morris, MD, Principal Investigator — University of Kentucky
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No